CLINICAL TRIAL: NCT05598333
Title: A Phase 2, Adaptive, Double-blinded, Placebo Controlled, Randomized, Multi-center Trial to Evaluate the Efficacy, Safety and Tolerability of Intracoronary Infusion of AB-1002 in Adult Subjects With New York Heart Association (NYHA) Class III Heart Failure and Non-ischemic Cardiomyopathy
Brief Title: Phosphatase Inhibition by Intracoronary Gene Therapy in Subjects With Non-Ischemic NYHA Class III Heart Failure
Acronym: GenePHIT
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AskBio Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ASK-CHF2-CS201
Record Dates: First submitted 2022-10-25; First posted 2022-10-28 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Congestive Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Genetic Therapy

STUDY DESIGN:
Intervention Model Description: Adaptive, double blinded, placebo controlled, randomized
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The IWRS will be programmed with blind-breaking instructions. In case of an emergency, the investigator has the responsibility for determining if unblinding of a subject's intervention assignment is warranted. If the investigator is unavailable, and a treating physician not associated with the study requests emergency unblinding, the emergency unblinding requests are forwarded to the emergency medical advice 24 hours/7 day service.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Treatment Group 1 AB-1002 (Experimental): Randomized in 1:1:1 into one of three groups. Group 1: 7.15E13vg/subject (n=30-50)
  Interventions: Drug: AB-1002
- Treatment Group 2 AB-1002 (Experimental): Randomized in 1:1:1 into one of three groups.
  Group 2: 1.43E14vg/subject (n=30-50)
  Interventions: Drug: AB-1002
- Treatment Group 3 (Placebo Comparator): Randomized in 1:1:1 into one of three groups.
  Group 3: Placebo (n=30-50)
  Interventions: Drug: AB-1002

INTERVENTIONS:
Drug: AB-1002 — Intracoronary Infusion of AB-1002 or placebo
  Other Names: Gene Therapy; NAN-101

SUMMARY:
This is a Phase 2 adaptive, double-blinded, placebo-controlled, randomized, multi-center trial study to evaluate the safety and efficacy of a single dose of AB-1002, administered via antegrade intracoronary artery infusion, in males and females age >18 years with non-ischemic cardiomyopathy and NYHA Class III symptoms of HF.

Subjects will be randomized into one of three treatment groups in a 1:1:1

DETAILED DESCRIPTION:
Subjects will be randomized into one of three treatment groups in a 1:1:1 fashion to either 7.15E13vg (n=30-50), 1.43E14 (n=30-50) or placebo group (n=30-50).

Approximately 90 to 150 subjects will be randomly assigned to study intervention Placebo

Study duration until the primary analysis at 52 week will be approximately 37 months including 25 months of recruitment and 52-week Observation Period after dosing. Once all the subjects complete the 52 weeks Observation Period, the treatment groups will be unblinded and primary analysis performed. Study participation duration: The study will last 52 weeks from dosing, with another 4 years of long-term follow-up for a total of 5 years. During the 4 year long-term follow up sites will contact subjects twice a year for two years, then once a year for the remaining two years for safety, efficacy assessments, and survival

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be age ≥18 years of age, at the time of signing the informed consent.
2. Chronic non-ischemic cardiomyopathy
3. 15% ≤ LVEF ≤ 35% by transthoracic echocardiography (TTE) at screening
4. 6MWT >50 meters
5. Medically stable, NYHA Class III HF for a minimum of 4 weeks while on appropriate medical therapy (defined below) including, but not limited to:

   1. Beta blocker therapy and ACE inhibitor or angiotensin receptor blocker (ARB) or sacubitril/valsartan combination therapy (Entresto) for ≥ 90 days prior to enrollment.

      May also receive aldosterone antagonist therapy. Doses of the above medications must be stable for ≥ 30 days prior to enrollment; and
   2. Cardiac resynchronization therapy (Zareba et al 2011), if clinically indicated, must have been implanted ≥ 90 days prior to enrollment. Internal cardioverter defibrillator (ICD) must be implanted, if clinically indicated ≥ 30 days prior to enrollment.
6. Women of childbearing potential must use at least one of the following acceptable birth control methods throughout the study and for 6 months after IP administration:

   * Surgically sterile (bilateral tubal ligation, hysterectomy, bilateral oophorectomy) 6 months minimum prior to IP administration
   * Intrauterine device in place for at least 90 days prior to receiving IP
   * Barrier methods (diaphragm plus spermicide or condom) starting at least 30 days prior to receiving IP
   * Abstinence (the subject must be willing to remain abstinent from screening to 6 months after receiving IP). Females are allowed to claim abstinence as their method of contraception only when it is the preferred and usual lifestyle of the subject
   * Surgical sterilization of the partner(s) (vasectomy) for >180 days prior to IP administration
   * Hormonal contraceptives starting > 90 days prior to IP. If hormonal contraceptives are started less than 90 days prior to receiving IP, subjects must agree to use a barrier method (diaphragm plus spermicide or condom) from screening through 90 days after initiation of hormonal contraceptives
7. Males subjects capable of fathering a child:

   * Must agree to use a condom and should also be advised of the benefit for a female partner to use a highly effective method of contraception as a condom may break or leak when having sexual intercourse with a woman of childbearing potential who is not currently pregnant from IP administration through 6 months after the time of IP administration
   * Must agree not to donate sperm for 6 months after time of receiving IP
   * Documented evidence of vasectomy in males for 180 days minimum prior to receiving IP is an acceptable form of contraception
   * Males who claim abstinence as their method of contraception are allowed, provided they agree to use barrier methods should they become sexually active from screening through 6 months after receiving IP. Males are allowed to claim abstinence as their method of contraception only when it is the preferred and usual lifestyle of the subject
8. Appropriate candidate for protocol-specified intracoronary infusion in the judgment of the infusing interventional cardiologist

   Exclusion Criteria:

   Subjects are excluded from the study if any of the following criteria apply:
9. Chronic ischemic cardiomyopathy secondary to obstructive coronary artery disease
10. Intravenous (IV) inotropic therapy, intra-aortic balloon pump (IABP) or percutaneous cardiac assist device therapy within 30 days prior to enrollment
11. Restrictive cardiomyopathy, obstructive cardiomyopathy, pericardial disease, amyloidosis, infiltrative cardiomyopathy, uncorrected thyroid disease, or dyskinetic LV aneurysm
12. Cardiac surgery or percutaneous coronary intervention (PCI) within 30 days prior to screening
13. Uncorrected Third degree heart block
14. Clinically significant myocardial infarction (MI) in the judgment of the subject's physician (e.g., ST elevation MI [STEMI] or large non-STEMI) within 6 months prior to enrollment
15. Prior heart transplantation, left ventricular reduction surgery (LVRS), cardiomyoplasty, passive restraint device (e.g., CorCap™ Cardiac Support Device), surgically implanted LVAD or cardiac shunt
16. Likely to receive cardiac resynchronization therapy, cardiomyoplasty, LV reduction surgery, heart transplant, conventional revascularization procedure, or valvular repair within 3 months of IP dosing in judgement of investigator.
17. Known hypersensitivity to contrast dyes (not easily controlled by antihistamines) used for angiography; history of, or likely need for, high-dose steroid pretreatment prior to contrast angiography.
18. Expected survival < 1 year in the judgment of the investigator
19. Active or suspected infection within 48 hours prior to intra-coronary infusion as evidenced by fever or positive culture
20. Known intrinsic liver disease (e.g., cirrhosis, hepatitis A, chronic hepatitis B or hepatitis C virus infection). If serology is positive and PCR is known to be negative, subject may be eligible (confirm with medical monitor).
21. Liver function tests (alanine aminotransferase [ALT], aspartate aminotransferase [AST], alkaline phosphatase) > 2x upper limit of normal (ULN) within 30 days prior to enrollment.
22. Chronic Kidney Disease Stage 5, dialysis dependent or eGFR<15 within 30 days prior to enrollment
23. Bleeding diathesis or thrombocytopenia defined as platelets <50,000 platelets/μL within 30 days prior to enrollment
24. Anemia defined as hemoglobin <10 g/dL or transfusion dependent within 30 days prior to enrollment
25. Neutropenia defined as absolute neutrophils <1500 mm3 within 30 days prior to enrollment
26. Known AIDS or HIV-positive status, or a previous diagnosis of immunodeficiency with an absolute neutrophil count <1000 cells/mm3
27. Previous participation in a study of gene transfer
28. Receiving investigational intervention or participating in another clinical study within 30 days of another investigational drug administration prior to administration of AB-1002 that may impact the therapeutic potential of AB-1002.
29. Pregnancy or breastfeeding or plans to become pregnant within the next 12 months at the time of screening
30. Subjects with any other condition which in the opinion of the investigator would preclude participation in the study (including risk for non-compliance and any intercurrent conditions that pose an undue medical hazard, or which could interfere with the interpretation of the study results)
31. Malignant neoplasm within 5 years of dosing, with the exception of those with negligible risk of metastasis or death (such as adequately treated carcinoma in situs of the cervix, basal or squamous cell skin cancer, localized prostate cancer or ductal carcinoma in situ)
32. Any documented history of non-compliance with medications, illicit drug use or laboratory evidence of illicit drug use during screen period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-10-20 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular Related Death | 52 weeks
NYHA Classification | 52 weeks
  NYHA Classification Change from baseline
Left Ventricular Ejection Fraction | 52 weeks
  LVEF change from baseline
Six Minute Walk Test | 52 weeks
  6MWT distance change from baseline

SECONDARY OUTCOMES:
Heart Failure Related Hospitalizations | 52 weeks
  Number of hospitalizations attributed to heart failure

CONTACTS AND LOCATIONS:
Locations (96):
- United States (37):
  - Cardiology P.C. Birmingham, Birmingham, Alabama
  - University of Arizona Sarvor Heart Center, Tucson, Arizona
  - University of California Irvine Medical Center, Irvine, California
  - University of California San Diego, La Jolla, California
  - University of California San Francisco, San Francisco, California
  - Baycare Medical Group, Clearwater, Florida
  - University of Miami, Coral Gables, Florida
  - University of Florida, Gainesville, Florida
  - Augusta University, Augusta, Georgia
  - Loyola Medicine Burr Ridge, Oakbrook Terrace, Illinois
  - University of Iowa, Iowa City, Iowa
  - University of Kansas Medical Center (KUMC), Kansas City, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - Mayo Clinic - Minnesota, Rochester, Minnesota
  - Aurora Saint Luke's Health System, Kansas City, Missouri
  - St. Louis University, St Louis, Missouri
  - Renown Health, Reno, Nevada
  - Morristown Medical Center - Cardiology, Morristown, New Jersey
  - Mt. Sinai New York, New York, New York
  - Stony Brook, Stony Brook, New York
  - Montefiore Medical Center, The Bronx, New York
  - Duke University, Durham, North Carolina
  - The Christ Hospital / The Linder Center for Research, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - LVH Cardiology, Allentown, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Medical University of South Carolina (MUSC) Medical Center, Charleston, South Carolina
  - Stern Cardiovascular, Germantown, Tennessee
  - Baylor Scott & White Advanced Heart Failure Clinic - Dallas, Dallas, Texas
  - Baylor College of Medicine (BCM) - Baylor Heart Clinic, Houston, Texas
  - Houston Methodist Debakey Cardiology Associates, Houston, Texas
  - University of Washington, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin
- Austria (4):
  - Medizinische Universität Graz, Graz
  - Kardiologie & Intensivmedizin Campus III, Linz
  - SALK University Hospital, Salzburg
  - NÖ Landesgesundheitsagentur, Sankt Pölten
- UZ Antwerpen, Edegem, Belgium
- Bulgaria (8):
  - Multiprofile Hospital for Active Treatment Sveti Georgi OOD, Pernik
  - Specialized Hospital For Active Cardiology Treatment Medica Kor EAD, Rousse
  - Multiprofile Hospital for Active Treatment "South West Hospital" OOD, Sandanski
  - Multiprofile Hospital for Active Treatment 'National Cardiology Hospital' EAD, Sofia
  - Acibadem City Clinic University Multiprofile Hospital For Active Treatment Tokuda EAD, Sofia
  - University Multiprofile Hospital for Active Treatment 'Sveta Ekaterina' EAD, Sofia
  - University Multiprofile Hospital for Active Treatment and Emergency Medicine N. I. Pirogov EAD, Sofia
  - University Multiprofile Hospital For Active Treatment Sofiamed OOD, Sofia
- Canada (10):
  - St. Boniface Hospital, Winnipeg, Manitoba
  - Memorial University Hospital, St. John's, Newfoundland and Labrador
  - London Health Sciences Centre, London, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - CIUSSS Saguenay Lac-St-Jean, Chicoutimi, Quebec
  - Institut de Cardiologie de Montréal, Montreal, Quebec
  - Centre Hospitalier de l'Université de Montréal - CHUM, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - CHU de Québec - Université Laval, Québec, Quebec
  - Institut Universitaire de Cardiologie et de Pneumologie de Québec - IUCPQ, Québec, Quebec
- Germany (6):
  - Technical University of Munich (TUM), München, Bavaria
  - Charité Universitaetsmedizin, Berlin
  - Universitaetsklinikum Freiburg | Herz-Zentrum Bad Krozingen (Heart Centre Bad Krozingen), Freiburg im Breisgau
  - Medizinische Hochschule Hannover (MHH), Hanover
  - Heidelberg University Hospital, Heidelberg
  - Universitätsklinikum Schleswig-Holstein, Kiel
- Hungary (6):
  - Semmelweis Egyetem, Varosmajori Sziv- és Ergyogyaszati Klinika, Budapest
  - Észak-Pesti Centrumkórház - Honvédkórház, Budapest
  - Budapesti Uzsoki Utcai Korhaz, Budapest
  - Somogy Varmegyei Kaposi Mor Oktato Korhaz - Kardiologiai Osztaly, Kaposvár
  - Pecsi Tudomanyegyetem Klinikai Kozpont, Szivgyogyaszati Klinika, Pécs
  - Szegedi Tudományegyetem, Szent-Györgyi Albert Klinikai Központ - Belgyógyászati Klinika, Szeged
- Netherlands (4):
  - Amsterdam UMC - Locatie AMC (Academisch Medisch Centrum), Amsterdam, North Holland
  - Radboud University Medical Center, Nijmegen
  - Erasmus Medisch Centrum, Rotterdam
  - Universitair Medisch Centrum (UMC) Utrecht, Utrecht
- Poland (3):
  - American Heart of Poland S.A. - MCSN, PAKS w Chrzanowie, Chrzanów
  - 1 Wojskowy Szpital Kliniczny z Poliklinika SPZOZ w Lublinie, Lublin
  - Uniwersytecki Szpital Kliniczny (USK) Nr 4 w Lublinie, Lublin
- Romania (6):
  - Spitalul Clinic Judetean De Urgenta Targu Mures, Târgu Mureş, County Mures
  - Spitalul Clinic Judetean De Urgenta Brasov- Sectia Cardiologie 3, Brasov
  - Spitalul Universitar de Urgenta Militar Central "Dr. Carol Davila", Sectia Clinica Cardiologie I, Bucharest
  - Spitalul Clinic Judetean De Urgenta Craiova- Sectia de Cardiologie, Craiova
  - Spitalul Universitar de Urgenta Bucuresti- Sectia Cardiologie 2, Târgu Mureş
  - Institutul De Boli Cardiovasculare Timisoara- Clinica de Cardiologie, Timișoara
- Spain (6):
  - Hospital Universitario de Bellvitge, Barcelona, Catalonia
  - Universidad de Navarra - Clinica Universidad de Navarra (CUN), Pamplona, Navarre
  - Hospital Ramon y Cajal | Cardiology - Research Unit, Madrid
  - Universidad Autonoma de Madrid (UAM) - Hospital Universitario La Paz (HULP), Madrid
  - Complejo Hospitalario Universitario Santiago de Compostela (CHUS), Santiago de Compostela
  - Hospital Clinico Universitario de Valencia (CHUV), Valencia
- United Kingdom (5):
  - Manchester Royal Infirmary, Manchester, Manchester
  - Leeds General Infirmary, Leeds, West Yorkshire
  - University Hospital of Wales, Cardiff
  - NHS Golden Jubilee, Glasgow
  - Imperial College London - National Heart & Lung Institute (NHLI) - Royal Brompton Campus, London

IPD SHARING:
Plan to Share IPD: No
No data will be shared with researchers outside of AskBio